CLINICAL TRIAL: NCT01198470
Title: A Prospective Clinical Investigation of the TRIUMPH Lumbar Disc: A Pilot Study
Brief Title: TRIUMPH Lumbar Artificial Disc IDE: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G090143
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Lumbar Degenerative Disc Disease
Keywords: Low back pain; Leg pain; Discogenic pain; Degenerative Disc Disease (DDD); Herniated disc; Radiculopathy
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain; Intervertebral Disc Displacement; Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRIUMPH® Artificial Disc (Experimental): Treatment of degenerative disc disease with the TRIUMPH Lumbar Artificial Disc. This is a non-randomized pilot study with only one arm (no control).
  Interventions: Device: TRIUMPH® Lumbar Artificial Disc

INTERVENTIONS:
Device: TRIUMPH® Lumbar Artificial Disc — The TRIUMPH® Lumbar Artificial Disc is an articulating artificial disc inserted using a posterolateral approach to the lumbar spine.

SUMMARY:
The purpose of this investigation is to evaluate the safety and effectiveness of the TRIUMPH® Lumbar Artificial Disc for the treatment of patients who are suffering from Degenerative Disc Disease (DDD) at one level from L1 to S1.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative Disc Disease in one vertebral level between L1 and S1
* Able to understand and sign informed consent
* Had at least 6 months of conservative treatment
* Oswestry Disability Index Score of at least 30 (one a 100 point scale)
* Other inclusion criteria as specified in approved IDE protocol

Exclusion Criteria:

* Bilateral leg pain
* Back or leg pain of unknown etiology
* Prior fusion surgery or another spinal device implanted at any other lumbar level
* Osteoporosis or osteopenia
* Other exclusion criteria as specified in approved IDE protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Health University Medical Center, Savannah, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRIUMPH® Artificial Disc
Started | 20
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | TRIUMPH® Artificial Disc
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Height [Mean (Standard Deviation); unit: inches] | 67.2 (3.0)
Weight [Mean (Standard Deviation); unit: pounds] | 178.1 (26.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change of at Least 15 Points in Pain/Disability Using the Oswestry Disability Index (ODI) Score at 24 Months Compared With the Score at Baseline
Description: The Oswestry Disability Index (ODI) is a commonly used outcome-measure questionnaire for low back pain in a hospital setting. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | TRIUMPH® Artificial Disc
Number analyzed (Participants) | 18
Participants | 16

2. Primary Outcome: Number of Participants With No Device Failures
Description: Any device requiring surgical revision, reoperation, removal or supplemental fixation will be considered a device failure
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | TRIUMPH® Artificial Disc
Number analyzed (Participants) | 20
Participants | 17

3. Primary Outcome: Number of Participants With Major Complications Defined as Major Vessel Injury or Neurological Damage
Description: Major vessel injury is defined as injury of the aorta or vena cava or other major vessels (e.g. iliac arteries, superior rectal artery, iliac veins, and their branches), caused by the surgery or device, resulting in significant blood loss or requiring additional surgery to correct. Neurological damage is defined as damage to the spinal cord or a nerve root caused by the surgery or device, resulting in neurologic deficit that persists for more than 3 months and is without improvement, is progressive, or involves motor loss. Major complications are reported on adverse event case report forms.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | TRIUMPH® Artificial Disc
Number analyzed (Participants) | 18
Participants | 0

4. Primary Outcome: Number of Participants Determined to Have a Normal Neurological Status
Description: Neurological status was assessed using a neurological status scale, which is based on four types of measurement parameters: motor, sensory, reflexes, and straight leg raise. The method for summarizing neurological status is described below. Each parameter (i.e. motor, sensory, reflexes, straight leg raise) is coded as follows:
  Motor 0 Total Paralysis
  1. Palpable or Visible Contraction
  2. Active Movement, Gravity Eliminated
  3. Active Movement, Against Gravity
  4. Active Movement, Against Some Resistance
  5. Active Movement, Against Full Resistance
  Sensory 0 Absent
  1. Impaired
  2. Normal
  Reflexes 0 Absent or Trace
  1. Hyper-reflexive
  2. Normal or hypo-reflexive
  Straight Leg Raise 0 0° - 70° (Abnormal)
  1 > 70°-90° (Normal)
  If all evaluations for the parameter are determined to be normal, then the parameter is given a normal status. If any evaluations for the parameter are abnormal, then the parameter is given an abnormal status.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | TRIUMPH® Artificial Disc
Number analyzed (Participants) | 18
Participants | 15

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | TRIUMPH® Artificial Disc
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRIUMPH® Artificial Disc (N=20)
Surgery - Index Level (Surgical and medical procedures) | 3 (3)
Gastric bypass to convert Lap Band (Gastrointestinal disorders) | 1 (1)
Headache and fatigue (General disorders) | 1 (1)
Intrauterine Growth Restriction (Renal and urinary disorders) | 1 (1)
Trauma (General disorders) | 1 (2)
Device migration (General disorders) | 1 (1)
Dural tear (General disorders) | 1 (1)
Dysesthesia - lower extremities (General disorders) | 1 (1)
Other (General disorders) | 1 (1)
Pain - back (General disorders) | 1 (1)
Weakness in bilateral legs (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRIUMPH® Artificial Disc (N=20)
Trauma (General disorders) | 6 (10)
Hypertension (Cardiac disorders) | 1 (1)
Dural tear (General disorders) | 1 (1)
Headache (General disorders) | 4 (4)
Pain - back (General disorders) | 4 (5)
Pain - back and hip (General disorders) | 2 (2)
Pain - back and lower extremities (General disorders) | 1 (1)
Pain - hip (General disorders) | 1 (1)
Pain - lower extremities (General disorders) | 3 (5)
Pain - lower extremities with dysesthesia (General disorders) | 1 (2)
Pain - neck and/or upper extremities (General disorders) | 3 (3)
Wound issue (General disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure type incidents (General disorders) | 1 (1)
Other (General disorders) | 6 (6)
Dysesthesia - lower extremities (General disorders) | 1 (1)
Paresthesia - lower extremities (General disorders) | 2 (2)
Urogenital (Renal and urinary disorders) | 1 (1)
Weakness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To prevent premature disclosure of trade secrets or other confidential information, PI agrees not to present, publish, or disclose study results or information about the investigational device without the express written consent of the sponsor.